CLINICAL TRIAL: NCT03450564
Title: The Effect of Community-Based Interventions on Increasing Family Planning Utilization in Pastoralist Community of Afar Region Ethiopia: A Cluster Randomized Controlled Trial
Brief Title: Effect of Community-Based Interventions on Increasing Family Planning Utilization in Pastoralist Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mekelle University (Other)
Responsible Party: Principal Investigator, Mussie Alemayehu, Principal Investigator, Mekelle University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Mekelle University RIF Project
Record Dates: First submitted 2017-08-10; First posted 2018-03-01 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Family Size
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The cluster randomized controlled trail will be designed to enhance family planning (FP) utilization in pastoralist community. An integrated behavioral model was used to guide the intervention. It has three arm and these are two community-based intervention and one control group and it was carried out for 9 months. Baseline and end line data was collected. The package of health education message was given to the married women of both arm (women and male involvement) arm and men in the male arm. Different modality was used in the men and women arm. These are involving faema leader, use of audiovisual materials of role model person in the community and providing training for health extension workers (HEW) and health care provider to assist for the faema leader.
Who Masked: Participant
Masking Description: The study was masked to the participants in which they don't disclose the type of intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Women Education (Experimental): In the married women arm there was an intervention with health education provision based on the baseline finding so as to fill the gap.Faema leader and video from (role model women who start to use FP, FP experts was used.Health extension workers were responsible in assisting the faema leader. Twice a month there was a provision of health education message about family planning for a total of 9 months.
  Interventions: Behavioral: Women Education
- Male Involvement (Experimental): In the married women arm there was an intervention with health education provision based on the baseline finding so as to fill the gap.Faema leader and video from (role model women who start to use FP, model who allows his wife to use FP, religious leader, FP experts was used.Health extension workers were responsible in assisting the faema leader. Twice a month there was a provision of health education message about family planning for a total of 9 months.
  Interventions: Behavioral: Male Involvement
- Control group (Other): The third arm in this community-based intervention was following the community without provision of male and married women education. In this arm, there was no intervention by the researchers. However, the activities performed by the government about family planning provision was maintained.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Women Education — This intervention intends to provide health education message for women enhance FP utilization in pastoralist community. It was cognizant that, Ethiopia is the second most populous country in Africa. And there is a great discrepancy between contraceptive use, unmet need for FP and maternal and child morbidity and mortality between the pastoralist and agrarian community. Pastoralist community in the country expressed as low contraceptive users, a high unmet need for FP and highest maternal and child morbidity and mortality. The previous study indicates that only 5.4% of the women use contraceptive. The most common reason mentioned for not using of contraceptive are lack of awareness, demand for a large number of children and male dominance in all decision making power in general and FP in particular. In light of this, the study hypothesized that working with men and educating women towards the use of FP could enhance the use of family planning utilization.
  Other Names: Women empowerment
  Arms: Women Education
Behavioral: Male Involvement — Male involvement was a feature of intervention in this arm. Comprehensive health education about FP was given in addition to the video message about FP. In pastoralist community the most reason mentioned for not using of FP are husband objection and religion influence. And most of the decisions are in the palm of husband to seek care for reproductive, maternal and neonatal health in general and FP in particular. Besides, the pastoralist community manifested by high total fertility rate and maternal and child morbidity and mortality.
  Other Names: women empowerment through men involvement
  Arms: Male Involvement
Other: Control group — The third group in this community based intervention was following the community without provision of male iand married women education. In this group there was no intervention by the researchers. However, the activities performed by the government about family planning provision was maintained.
  Other Names: Active comparator
  Arms: Control group

SUMMARY:
The cluster randomized controlled trial was done in Pastoralist community of Afar region, Ethiopia for a total of nine months. There was three arms in the study. The type of randomization will be a cluster randomized controlled trial where kebele are randomized to two different interventions and control groups. These interventions are women education to use family planning and male education/involvement to enhance family planning use in the community.

DETAILED DESCRIPTION:
The study hypothesized that doing on women education and men education/involvement in family planning utilization would be a practical way to achieve for an increment of family planning utilization in Pastoralist community of Afar region. The study was carried out in Afar region, North Eastern Ethiopia from Jan1, 2018, to September 5, 2018. A three-arm, parallel randomized controlled trial was used to answer the objective of the study. The type of randomization will be a cluster randomized controlled trial where kebele are randomized to two different interventions and one control groups together. These interventions are women education to use family planning and male education/involvement to enhance family planning use in the community.

The unit of randomization was clustered which are kebeles in a different districts. From a given district 11 Kebele were selected randomly gives a total of 33 kebele. The 33 cluster were allocated to the 2 interventions and one control arms. The detail description of the two interventions and one control arm is described below.

* Arm 1): existing standard family planning service provision by the government health sectors.
* Arm 2): It focuses on the involvement of men to enhance the utilization of family planning by their wives and educating the women in the male intervention area.
* Arm 3): It deals with educating married women to use family planning.

Data collection tool, procedures, and follow-up We develop the quantitative tool based on the previous finding in the region. It contains baseline and end line data collection with a nine-month duration. The tool was piloted on 10% (118) of the sample and it was tested for reliability and validity test for items of of knowledge, attitude, subjective norm, perceived behavioral control over FP use, intention to use for FP and male involvement. Accordingly, modification was made based on the finding of reliability and validity test. A tool which has a All items were subjected to exploratory factor analysis to identify the relevant constructs. Items with low load factor (less than 0.3) to the identified constructs were deleted. Then the reliability test was done to assess the consistency of items in each construct (Cronbach's Alpha > 0.7). At the end, a final tool was prepared based on the finding of the reliability and validity test. Then, it was pretested in 5% (45) of the sample. 6 clinical nurse data collectors and 2 supervisors were used to collect the data after they got training on the items and how to use mobile based application. They were assigned to a different cluster of a given district. The data was collected using mobile based application called open data kit (ODK) for a one month. A similar procedure was used in the end line data collection. Immediately after the data checked for its completeness, it was sent to the Mekelle University (MU) Server. Hence, at the middle of the intervention, qualitative data was collected to identify the participants acceptability and documenting best experience of the intervention.

Intervention description:

The community-based intervention in this study includes two components. These are educating women to use family planning and male involvement for use of family planning.

Analysis plan and statistics methods The type of data used in the intervention study was a repeated cross-sectional. The data collected using ODK, was exported to R software version 3.4.2 for analysis.Intention to treat analysis was used as a framework of analysis. All the analysis was used with 95% confidence interval and p-value <0.05 to declared statistically significant. Since the number of clusters per arm was 11, a cluster level summary was used to compare the control group with the intervention (women education and male involvement). A separate cluster level summaries analysis was done for control Vs the women arm and control with the male arm by considering the effect of cluster. Finally, the result was described with t-test, df, P-value, mean value of both group and 95% CI of the adjusted risk. Moreover, prevalence ratio of the end line FP user over the baseline FP was done.

Ethical consideration Permission to undertake the study was obtained from Mekelle University College of Health Sciences institutional review board with a reference number ERC 1435/2018. And an official letter of cooperation was given to Afar Regional Health Bureau. Permission was obtained from all relevant authorities in the Afar regional health bureau and participating district health offices (Afambo, Kori and Mille). At the beginning community consent was secured from the influential group (religious and clan leader). Verbal consent was secured before conducting interviews and parental/guardian consent was waived to include the minors to the study by the ethical board. The informed consent was secured continuously every three months. A one-page consent letter was attached to the cover page of each questionnaire as an information sheet which includes a detail description about the benefit and risk of participating in the study, participation is on voluntary basis, the right to withdraw from the study, identification of informant was possible only through specific identification numbers and the privacy of collected information. Data collection was conducted through electronically smartphone mobile based application (ODK) and it was confidentially.

ELIGIBILITY:
Inclusion Criteria:

* A household was considered eligible for the study if the following criteria are met:

  * at least one married women with reproductive age group (15-49) year's child
  * able to provide a consent and voluntary to participate in the study
  * Cluster which has more than 30 married women. A household was excluded if the woman or her husband will not volunteer to participate in the study.

Exclusion Criteria:

* Married women who are not volunteer to provide informed consent
* Married women who are declared infertile

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 891 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Family planning utilization | 9 months
  the family planning utilization will be assessed by asking the participant either use or not use of contraceptive during data collection.Both the ever use or current use of the family planning will be collected from the married women.

SECONDARY OUTCOMES:
Intention to use family planning | 9 months
  A total of 9 items which has a natural ascending order was used. The items includes the following points. I am not clear with the benefits of using family planning , at this moment, I can list some of the benefits of family planning use I would gain if I use it, I am happy if I could use family planning to space the number of children I would have in the future, I am willing to use family planning to space/limit number of children, I have already decided that I should use family planning in the near future, I have ever used family planning in the previous 6 months and I found it relevant me, I have ever used FP in the past 6 months and I am quite sure I will continue using it in the future and It is expected that women in our community should use family planning and so do I.

CONTACTS AND LOCATIONS:
Overall Officials: Belete Assefa, Study Director — Mekelle University College of Health Science, Academic and research Director; Mohamed Ahmed, Study Chair — Semera University, Director of Research and community Service; Yasin Habib, Study Chair — Deputy Head of Afar regional Health Bureau; Mussie Alemayehu, Principal Investigator — Mekelle University, College of Health Sciences, School of Public Health
Locations (1):
- Afar Region, Semera, Zone 1, Ethiopia

IPD SHARING:
Plan to Share IPD: No
The individual data will not be shred to other individual to keep the confidentiality of the study.

REFERENCES:
- [Background] Alemayehu et al. Family planning use and associated factors among pastoralist community of afar region, eastern Ethiopia. BMC Women's Health (2016) 16:39 DOI 10.1186/s12905-016-0321-7 Afework B., Alemayehu M., Znabu H., Araya AM., Mohammed A., Afework M. Factors influencing contraceptive use among women of reproductive age from the pastoralist communities of Afar, Ethiopia: a community-based cross-sectional study. Ethiop. J. Health Dev. 2018;32(Special Issue):28-33 Znabu H., Alemayehu M, Araya AM., Afework M. Drivers to have more children in the pastoralist communities of Afar, Ethiopia: an explorative qualitative study. Ethiop. J. Health Dev. 2018;32(Special Issue):21-27 Alemayehu M., Araya AM., Afework M.A review of evidence on barriers to and facilitators of the utilization of reproductive, maternal and neonatal health services among pastoralist communities in Sub-Saharan Africa. Ethiop. J. Health Dev. 2018;32(Special Issue):43-49 Key CW., Araya AM.,Mark S., Mussie A.,Selemawit AB.,Abiy HS.,Ephrem TL., Afework M.Best practices for addressing socio-cultural barriers to reproductive, maternal and neonatal health service utilization among women from pastoralist communities of Afar, Ethiopia: A qualitative study. [Ethiop. J. Health Dev. 2018;32(Special Issue):4-12 Alemayehu M.,Araya AM, Kibrom B, Yemane G., Tesfay H.,Selemawit AB., Mohammed A., Afework M.The Levels of utilization of reproductive, maternal and neonatal health services among women from pastoralist communities in Afar, Ethiopia: across-sectional survey. Ethiop. J. Health Dev.2018;32(Special Issue):34-42
- [Derived] Alemayehu M, Medhanyie AA, Reed E, Kahsay ZH, Kalayu M, Mulugeta A. Effects of continuum of care for maternal health service utilisation on intention to use family planning among pastoralist women of Ethiopia: a robust regression analysis and propensity score matching modelling. BMJ Open. 2023 Jul 12;13(7):e072179. doi: 10.1136/bmjopen-2023-072179. PMID 37438064
- [Derived] Alemayehu M, Medhanyie AA, Reed E, Bezabih AM. Use of community-based interventions to promote family planning use among pastoralist women in Ethiopia: cluster randomized controlled trial. BMC Womens Health. 2021 Aug 18;21(1):305. doi: 10.1186/s12905-021-01434-x. PMID 34407805
- [Derived] Alemayehu M, Medhanyie AA, Reed E, Mulugeta A. Individual-level and community-level factors associated with the family planning use among pastoralist community of Ethiopia: a community-based cross-sectional study. BMJ Open. 2020 Sep 9;10(9):e036519. doi: 10.1136/bmjopen-2019-036519. PMID 32907899